CLINICAL TRIAL: NCT00386126
Title: Randomized Trial to Assess the Effects of Iron Supplementation in Heart Failure Patients With Anemia: The IRON-HF Study
Brief Title: Iron Supplementation in Heart Failure Patients With Anemia: The IRON-HF Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCPA 06-115
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-08

CONDITIONS: Heart Failure; Anemia
Keywords: Heart Failure; Anemia; Treatment
MeSH Terms: conditions — Heart Failure; Anemia | interventions — WW Domain-Containing Oxidoreductase; ferrous sulfate

INTERVENTIONS:
Drug: Iron Sucrose IV 200mg, once a week, for 5 weeks
Drug: Ferrous sulfate 200mg PO TID, for 8 weeks

SUMMARY:
Anemia has been demonstrated to be a common finding in patients with heart failure (HF). Previous studies in hospitalized patients with HF have found a prevalence of anemia ranging from 15% to 63%. More importantly, anemic patients with HF have increased morbidity and mortality. The mechanisms underlying anemia in HF are multifactorial, involving mild to moderate forms of anemia of chronic disease and ferropenic anemia. The clinical impact of iron supplementation in HF patients who have a relatively preserved renal function and either chronic disease anemia, ferropenic anemia or both remains largely unknown. The route of iron administration that could be most clinically effective is also unclear. Thus, the primary aim of the IRON-HF study is to assess the effects of iron supplementation alone (IV or PO) on parameters of functional capacity in HF patients with anemia with decreased availability of iron.

DETAILED DESCRIPTION:
The IRON-HF study is an investigator initiated, multicenter, prospectively designed,randomized, double-blind, placebo controlled clinical trial.

Randomization:Each of the eight participating centers will randomize patients by telephone contact with the randomization center at Hospital de Clínicas de Porto Alegre. The randomization system will be based on a computerized table of random numbers and performed in blocks of three per participating center.

Blinding:Each participating center will elect a third party blind individual (usually a RN) who will open the allocated medication box, prepare iron sucrose infusions or saline and administer to patients in opaque devices. Both patient and attending physicians and/or nurses will be blind to allocated therapy. Oral medications and oral placebo will be identical in all aspects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Outpatients followed at a HF Clinic in a tertiary care Hospital with clinical diagnosis of HF for at least 3 months before study entry;
* NYHA functional class II to IV, who are able to perform ergospirometry;
* Documentation of LVEF < 40% within the last 6 months;
* Adequate baseline therapy for HF based on patient's functional class (β-blockers, ACE inhibitors irrespective of functional class except if contra-indications, digoxin, spironolactone if NYHA class III or IV);
* Stable baseline HF therapy with same doses of medications and no intent to increase doses for the following 3 months;
* Hemoglobin ≤ 12 g/dl and > 9 g/dl;
* Transferrin saturation < 20% and ferritin < 500 µg/L;
* Ability to provide written informed consent.

Exclusion Criteria:

* Any clinically overt bleeding: gastrointestinal bleeding, hypermenorrhea, history of peptic ulcer without evidence of healing or inflammatory intestinal diseases;
* Uncorrected hypothyroidism;
* Other inflammatory, neoplastic or infectious disease;
* Serum creatinine > 1,5 mg/dl;
* Previous intolerance to oral elemental iron compounds;
* HF due to alcoholic cardiomyopathy, current regular drinker of alcoholic beverages or HF due to peripartum cardiomyopathy;
* Recent admission for decompensated HF (last month)
* Recent myocardial revascularization procedures (last 3 months);
* Recent ACS, stroke or TIA (last 3 months);
* Active or metastatic neoplastic disease with life expectancy of less than a year;
* Patients in heart transplantation list;
* Patients that had participated in any other clinical trial or study within the last month;
* Pregnant or lactating women;
* Pre-menopausal women that are not using any effective method of contraception;
* Patients using prohibited medications or that have not yet accomplished the wash-out period;
* Patients currently participating in cardiovascular rehabilitation programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117
Dates: Start 2006-08

PRIMARY OUTCOMES:
The primary endpoint of the IRON-HF study is to assess the impact of iron supplementation alone (IV or PO) on changes in oxygen maximal consumption (peak VO2) assessed by ergospirometry over a 3-month follow-up period.

SECONDARY OUTCOMES:
New York Heart Association (NYHA) functional class
BNP (B-type natriuretic peptide) levels
Quality of life using the Living with Heart Failure Minnesota Questionnaire
Left ventricular ejection fraction (LVEF) as assessed by the bi-planar modified Simpson method in two-dimensional echocardiography
Renal function as assessed by the serum levels of creatinine
Incidence of hospitalizations due to HF
Mortality
Incidence of adverse events (drug tolerance).

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Clausell, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Cardiovascular Division, Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Beck-da-Silva L, Piardi D, Soder S, Rohde LE, Pereira-Barretto AC, de Albuquerque D, Bocchi E, Vilas-Boas F, Moura LZ, Montera MW, Rassi S, Clausell N. IRON-HF study: a randomized trial to assess the effects of iron in heart failure patients with anemia. Int J Cardiol. 2013 Oct 9;168(4):3439-42. doi: 10.1016/j.ijcard.2013.04.181. Epub 2013 May 13. PMID 23680589